CLINICAL TRIAL: NCT04019483
Title: Improved Prediction of Recurrent Stroke and Detection of Small Volume Stroke
Acronym: ENCLOSE
Status: Terminated | Type: Observational
Why Stopped: Insufficient inclusion and end of funding
Sponsor: UMC Utrecht (Other)
Collaborators: Dutch Heart Foundation (Other); Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Principal Investigator, Jan. W. Dankbaar, MD, PhD, Principal Investigator, UMC Utrecht
Other Study IDs: NL62233.041.17
Record Dates: First submitted 2019-07-10; First posted 2019-07-15 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Ischemic Stroke
Keywords: Recurrence; Infarct detection; CT; MRI; Diagnosis; Prognosis
MeSH Terms: conditions — Ischemic Stroke; Recurrence; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rationale: Over 20.000 people suffer an ischemic stroke in the Netherlands each year. Large artery occlusions are easy to identify and can be treated with endovascular clot removal. 70% of patient will however suffer from a more distal occlusion resulting in small volume stroke or a transient ischemic attack (TIA). Small ischemic lesions are hard to detect with current acute stroke protocols. TIA and small volume stroke patients, are at an increased risk for recurrent stroke, making immediate diagnosis critical. Because thrombo-embolic sources often cause these strokes, identifying and treating the underlying aetiology has the potential to radically lower the risk of recurrence and improve the outcome of these patients.

Objectives: 1) To identify clinical and imaging predictors of recurrent stroke; 2) To improve early detection of small volume stroke with admission computed tomography perfusion (CTP) in patients with suspected acute ischemic stroke with small volume stroke or no ischemia on admission imaging.

Study design: Prospective, multicenter cohort study.

Study population: All patients who visited the University Medical Center (UMC) Utrecht, the Amsterdam University Medical Centers (Amsterdam UMC), location Academic Medical Center (AMC) or the St. Antonius Hospital and who underwent a CT-scan of the brain within 9 hours after onset of stroke symptoms with an age ≥18 years. Within 36 months, 720 patients will be enrolled in the study. Of these patients, 300 patients will be included for the follow-up magnetic resonance imaging (MRI).

Main study parameters/endpoints: The main study endpoints are: 1) Stroke recurrence rate at 2 years; 2) Presence and volume of acute ischemic lesions on follow-up diffusion weighted imaging MRI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Time from symptom onset until imaging is <9 hours*;
* Clinical diagnosis of acute ischemic stroke or TIA;
* Informed consent from patient or family after the admission scan (unless the patient died).

  * Patients who awaken with stroke symptoms can only be included if they went to sleep without any stroke symptoms and the time from going to sleep until imaging is less than 9 hours.

Exclusion Criteria:

* Patients with another diagnosis such as intracerebral hemorrhage, subarachnoid hemorrhage or tumor;
* Patients with known contrast allergy or renal failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years or older with acute stroke symptoms who visited the UMC Utrecht, the Amsterdam UMC, location AMC or the St. Antonius Hospital and who underwent a CT-scan within 9 hours after onset of stroke symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 439 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Recurrent ischemic stroke | 2 years

SECONDARY OUTCOMES:
Recurrent ischemic stroke | 90 days
modified Rankin scale | 90 days
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6 with "0" being perfect health without symptoms to "6" being death.
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
  9 - No data.

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Amsterdam UMC, location AMC, Amsterdam, North Holland
  - St. Antonius Hospital, Nieuwegein, Utrecht
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kauw F, Velthuis BK, Takx RAP, Guglielmo M, Cramer MJ, van Ommen F, Bos A, Bennink E, Kappelle LJ, de Jong HWAM, Dankbaar JW. Detection of Cardioembolic Sources With Nongated Cardiac Computed Tomography Angiography in Acute Stroke: Results From the ENCLOSE Study. Stroke. 2023 Mar;54(3):821-830. doi: 10.1161/STROKEAHA.122.041018. Epub 2023 Feb 13. PMID 36779342
- [Derived] Kauw F, van Ommen F, Bennink E, Cramer MJ, Kappelle LJ, Takx RA, Velthuis BK, Viergever MA, Wouter van Es H, Schonewille WJ, Coutinho JM, Majoie CB, Marquering HA, de Jong HW, Dankbaar JW. Early detection of small volume stroke and thromboembolic sources with computed tomography: Rationale and design of the ENCLOSE study. Eur Stroke J. 2020 Dec;5(4):432-440. doi: 10.1177/2396987320966420. Epub 2020 Oct 23. PMID 33598562